CLINICAL TRIAL: NCT06435455
Title: A Phase Ib/II Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of GH21 Capsule Combined With D-1553 Tablets in Patients With Locally Advanced or Metastatic Solid Tumors Harboring KRAS G12C Mutation
Brief Title: GH21 Combined With D-1553 in KRAS G12C Mutant Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Genhouse Bio Co., Ltd. (Other)
Collaborators: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH21C203
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Locally Advanced or Metastatic Solid Tumors Harboring KRAS G12C Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "GH21 + D-1553" Group (Experimental): GH21 capsules combined with D-1553 tablets were administrated orally
  Interventions: Drug: GH21; Drug: D-1553

INTERVENTIONS:
Drug: GH21 — GH21 Capsules, Oral Drug Specification: 3mg/capsule; 10mg/capsule
Drug: D-1553 — D-1553 Film-coated Tablets, Oral Drug Sepcification: 200mg/tablet

SUMMARY:
This s a multi-center, open-label phase Ib/II study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of GH21 combined with D-1553 in patients with advanced or metastatic solid tumors harboring KRAS G12C mutation.

DETAILED DESCRIPTION:
This study includes 2 parts: dose escalation(Phase Ib) and dose expansion (Phase II). The objective of the dose escalation part is to evaluate the safety, tolerability and pharmacokinetics of GH21 in combination with D-1553 in patients with advanced solid tumors harboring KRAS G12C mutation and to determine the RP2D for the combination therapy. In the dose expansion part, preliminary efficacy and safety of the combination therapy at the RP2D will be further explored in patients with specific cancer harboring KRAS G12C mutation.

ELIGIBILITY:
Inclusion Criteria:

* The patient or his legal representative is able to understand and voluntarily sign a written informed consent (before commencing this study and any research procedure);
* Age ≥18 years old, male or female;
* KRAS G12C mutant advanced solid tumor;
* ECOG Performance Status of 0 or 1
* At least one measurable lesion as defined by RECIST 1.1

Exclusion Criteria:

* acute myocardial infarction, unstable angina pectoris, coronary artery bypass grafting, cerebrovascular accident, or transient ischemic attack within 6 months before first administration; Grade III-IV heart failure based on the New York Heart Association Cardiac Function Scale at screening; During screening, echocardiography (ECHO) showed left ventricular ejection fraction (LVEF) ≤50%;
* Patients who have a history of severe allergy, or have a history of allergy to the experimental drug/any excipient/combination drug, or have a history of allergy to multiple drugs;
* There is an active infection (≥ grade 2) requiring anti-infective treatment or an unexplained fever exceeding 38 ° C within 28 days before the first dose;
* Any toxicity from previous antitumor therapy prior to initial administration has not returned to CTCAE 5.0 rating ≤ Class 1 (unless hair loss, grade 2 peripheral neuropathy, and/or other grade ≤2 adverse events that do not pose a safety risk);
* Pregnant and lactating women;
* The investigator considers that there are any clinical or laboratory abnormalities or other reasons to be unsuitable for participating in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicities Incidence Count Among Study | 2 years
  Incidence of dose limiting toxicities (DLTs) in the dose escalation phase.
Participants Number of Participants Reporting Adverse Events (AEs) or Serious Adverse Events (SAEs)Objective | 2 years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs , etc

SECONDARY OUTCOMES:
response rate (ORR) based on RECIST 1.1 criteria | 2 years
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR)
Duration of response (DOR) based on RECIST 1.1 criteria | 2 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) based on RECIST 1.1 criteria | 2 years
  DCR is defined as proportion of participants with complete response, partial response, stable disease(CR+PR+SD).
Progression-free survival (PFS) based on RECIST 1.1 criteria | 2 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first.
Overall survival (OS) | 2 years
  OS is defined as the interval of time between the date of first treatment until death, loss to follow up or termination of the study by the sponsor
Plasma concentration (Cmax) | 2 years
  Peak Plasma concentration
Time to achieve Cmax (Tmax) | 2 years
  Time to achieve Cmax
Area under the plasma concentration-time curve (AUC) | 2 years
  Area under the plasma concentration-time curve

IPD SHARING:
Plan to Share IPD: No